CLINICAL TRIAL: NCT02315027
Title: Intrathecal Autologous Mesenchymal Stem Cell Therapy in Multiple System Atrophy (MSA) - Effect of Dose and Natural History
Brief Title: Mesenchymal Stem Cell Therapy in Multiple System Atrophy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Wolfgang Singer, MD, Associate Professor, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12-005950; R01FD004789 (FDA); R01NS092625 (NIH)
Record Dates: First submitted 2014-10-31; First posted 2014-12-11 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: MSA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 1 dose of 1 × 10(7) MSCs (Experimental): Group 1: Participants will receive a single intrathecal dose of 1 × 10(7) mesenchymal stem cells (MSCs)
  Interventions: Biological: Autologous Mesenchymal Stem Cells
- 2 doses of 5 × 10(7) MSCs (Experimental): Group 2: Participants will receive one intrathecal dose of 5 × 10(7) mesenchymal stem cells (MSCs), followed by a second intrathecal dose of 5 × 10(7) MSCs approximately one month later
  Interventions: Biological: Autologous Mesenchymal Stem Cells
- 2 doses of 1 × 10(8) MSCs (Experimental): Group 3: Participants will receive one intrathecal dose of 1 × 10(8) mesenchymal stem cells (MSCs), followed by a second intrathecal dose of 1 × 10(8) MSCs approximately one month later
  Interventions: Biological: Autologous Mesenchymal Stem Cells
- 10 doses of 5 x 10(7) (±20%) MSCs (Experimental): Group 4: Participants will receive up to 10 doses of 5 x 10(7) (±20%) mesenchymal stem cells (MSCs) approximately 6 months apart.
  Interventions: Biological: Autologous Mesenchymal Stem Cells
- 10 doses of 2.5 x 10(7) (±20%) MSCs (Experimental): Group 5: Participants will receive up to 10 doses of 2.5 x 10(7) (±20%) mesenchymal stem cells (MSCs) approximately 6 months apart.
  Interventions: Biological: Autologous Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Autologous Mesenchymal Stem Cells — single dose of 1 × 10(7) cells intrathecally
  Arms: 1 dose of 1 × 10(7) MSCs
Biological: Autologous Mesenchymal Stem Cells — 2 doses of 5 × 10(7) cells intrathecally each 1 month (±4 days) apart
  Arms: 2 doses of 5 × 10(7) MSCs
Biological: Autologous Mesenchymal Stem Cells — 2 doses of 1 × 10(8) cells intrathecally each 1 month apart
  Arms: 2 doses of 1 × 10(8) MSCs
Biological: Autologous Mesenchymal Stem Cells — Ten doses of 5 x 10(7) (±20%) cells intrathecally six months (±1 month) apart
  Arms: 10 doses of 5 x 10(7) (±20%) MSCs
Biological: Autologous Mesenchymal Stem Cells — Ten doses of 2.5 x 10(7) (±20%) cells intrathecally six months (±1 month) apart
  Arms: 10 doses of 2.5 x 10(7) (±20%) MSCs

SUMMARY:
The purpose of this study is to determine whether mesenchymal stem cells (MSCs) can be safely delivered to the cerebrospinal fluid (CSF) of patients with multiple system atrophy (MSA). Funding Source - FDA OOPD.

DETAILED DESCRIPTION:
The primary aim is to evaluate the safety and tolerability of intrathecal injection of autologous MSCs in a dose escalation study in patients with MSA. Safety secondary goals include to monitor changes in peripheral blood and in components of CSF, and monitor for any changes of nervous system structures using MRI. Efficacy secondary goals include evaluating potential efficacy by providing a number of studies and instruments that will detect changes in the course of the disease in terms of autonomic and neurologic symptoms and deficits.

ELIGIBILITY:
Inclusion Criteria

1. Participants aged 30-80 years old with a diagnosis of MSA based on clinical criteria and standardized autonomic testing. This approach allows for identification of patients with MSA with very high specificity and is yet sensitive enough to allow for enrollment of patients at a disease stage at which an intervention on the natural disease course has a meaningful impact on patient outcome. Patients therefore have to fulfill Gilman Criteria (2000) for probable MSA of the parkinsonian subtype (MSA-P) or cerebellar subtype (MSA-C) and have findings on autonomic function testing suggestive of MSA (CASS ≥5 or a TST% ≥25%).
2. Participants who are less than 4 years from the time of documented MSA diagnosis.
3. Participants with an anticipated survival of at least 3 years in the opinion of the investigator.
4. Participants who are willing and able to give informed consent.
5. "Normal" cognition as assessed by Mini-Mental State Examination (MMSE). We will require a value >24.

Exclusion Criteria

Any of the following conditions will exclude the participant from entering the study:

1. Women of childbearing potential who do not practice an acceptable method of birth control. Acceptable methods of birth control in this study are: surgical sterilization, intrauterine devices, partner's vasectomy, a double-protection method (condom or diaphragm with spermicide), hormonal contraceptive drug (i.e., oral contraceptive, contraceptive patch, long-acting injectable contraceptive) with a required second mode of contraception.
2. Participants with a clinically significant or unstable medical or surgical condition that, in the opinion of the investigator, might preclude safe completion of the study or might affect the results of the study. These include conditions causing significant central nervous system (CNS) or autonomic dysfunction, including congestive heart failure, recent (<6 months) myocardial infarct, cardiopulmonary disease, severe, uncontrolled hypertension, thrombocytopenia (<50 x 10(9)/L), severe anemia (<8g/dl), immunocompromised state, liver or kidney disease (creatinine >2.3mg/dl), uncontrolled diabetes mellitus (HbA1c >10g%), alcoholism, amyloidosis, uncontrolled hypothyroidism, sympathectomy, unstable peripheral neuropathies, concurrent infections, orthopedic problems that compromise mobility and activity of daily living, cerebrovascular accidents, neurotoxin or neuroactive drug exposure, parkinsonism due to drugs (including neuroleptics, alpha-methyldopa, reserpine, metoclopramide).
3. Participants with malignant neoplasms.
4. Participants who have taken any investigational products within 60 days prior to baseline.
5. Medications that could affect autonomic function. If patients are taking those medications, those will be suspended prior to autonomic testing. Therapy with midodrine, anticholinergic, alpha and beta adrenergic antagonists or other medications that affect autonomic function will be withdrawn 48 hours prior to autonomic evaluations. Fludrocortisone doses up to 0.2 mg per day will be permitted.
6. Diseases with features of Parkinsons Disease; e.g., diffuse Lewy body disease, progressive supranuclear palsy, essential tremor, hereditary olivopontocerebellar atrophy, or postencephalitic parkinsonism.
7. Dementia (DSM-IV criteria - American Psychiatric Association 1994). The score on the Mini-Mental State Examination must be >24.
8. History of electroconvulsive therapy.
9. History of brain surgery for Parkinsons disease.
10. Patients with contraindication for MRI scanning, including those with MRI-incompatible pacemakers
11. Patients with active systemic infection or local infection, which is close to the spinal injection site

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Adverse event frequency (by severity, type, attribution, and intervention dose). | 14 months

SECONDARY OUTCOMES:
Rate of change of Unified Multiple System Atrophy Rating Scale (UMSARS) I score from baseline to 12 months (or last available date), compared with placebo limb of Rifampicin trial (historical control cohort). | 12 months
Rate of change from baseline to 12 months (or last available date) in UMSARS II score. | 12 months
Rate of change from baseline to 12 months (or last available date) in UMSARS total score. | 12 months
Rate of change in COMPASS-select score from baseline to 12 months. | 12 months
Change in CASS score and thermoregulatory sweat test (TST) % from baseline to 12 months. | 12 months
MRI morphometric changes using dedicated algorithms to evaluate rate of atrophy of defined areas of brain from baseline to 12 months. | 12 months
Change in CSF biomarkers from baseline to 2 months. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Singer, MD, Principal Investigator — Mayo Clinic; Phillip Low, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Camilleri ET, Gustafson MP, Dudakovic A, Riester SM, Garces CG, Paradise CR, Takai H, Karperien M, Cool S, Sampen HJ, Larson AN, Qu W, Smith J, Dietz AB, van Wijnen AJ. Identification and validation of multiple cell surface markers of clinical-grade adipose-derived mesenchymal stromal cells as novel release criteria for good manufacturing practice-compliant production. Stem Cell Res Ther. 2016 Aug 11;7(1):107. doi: 10.1186/s13287-016-0370-8. PMID 27515308